CLINICAL TRIAL: NCT06891066
Title: A Phase 2b, Randomized, Active-Controlled, Open-Label Clinical Study to Evaluate a Switch to Islatravir (ISL) and Ulonivirine (ULO) Once Weekly in Adults With HIV-1 Virologically Suppressed on Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) Once Daily
Brief Title: A Study of Islatravir (ISL) and Ulonivirine (ULO) Once Weekly (QW) in Virologically Suppressed Adults With Human Immunodeficiency Virus Type 1 (HIV-1) (MK-8591B-060)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8591B-060; MK-8591B-060 (Other: MSD)
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Human Immunodeficiency Virus Type 1 (HIV-1) Infection
Keywords: HIV-1
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — islatravir; ulonivirine; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ISL + ULO in Group 1 (Experimental): In part 1 of the study, participants will receive ISL 2mg + ULO 200mg orally once a week (QW) for 48 weeks. In part 2 (2nd 48 weeks), participants will continue to receive ISL 2mg + ULO 200mg once a week till week 96.
  Interventions: Drug: ISL; Drug: ULO
- BIC/FTC/TAF in Group 2 (Active Comparator): In part 1 of the study, participants will receive BIC 50mg/FTC 200mg/TAF 25mg orally once daily (QD) for 48 weeks.
  Interventions: Drug: BIC/FTC/TAF
- ISL + ULO in Group 2 (Experimental): In part 2 of the study, participants previously on BIC/FTC/TAF (for the 1st 48 weeks, or part 1) will switch to ISL + ULO, to week 96.
  Interventions: Drug: ISL; Drug: ULO

INTERVENTIONS:
Drug: ISL — ISL 1mg oral capsule will be administered as 2mg orally (each capsule 1mg) as part of ISL and ULO combination to group 1 participants for 96 weeks and for group 2 participants in part 2 of the study from 49 to 96 weeks.
  Other Names: MK-8591; Islatravir
  Arms: ISL + ULO in Group 1; ISL + ULO in Group 2
Drug: ULO — ULO 100mg oral tablet will be administered as 200mg (2 tablets) orally as part of ISL and ULO combination to group 1 participants for 96 weeks and for group 2 participants in part 2 of the study from 49 to 96 weeks.
  Other Names: MK-8507; Ulonivirine.
  Arms: ISL + ULO in Group 1; ISL + ULO in Group 2
Drug: BIC/FTC/TAF — BIC 50mg oral tablet/FTC 200mg oral tablet/TAF 25 mg oral tablet administered orally to group 2 participants for 48 weeks in part 1 of the study.
  Other Names: BIKTARVY®
  Arms: BIC/FTC/TAF in Group 2

SUMMARY:
Investigators are trying to find better treatments for people with HIV-1. In this clinical study, investigators want to see how well a new treatment called ISL+ULO, taken once a week, works compared to an existing treatment called BIC/FTC/TAF, which is taken every day. Investigators will check how many people still have a high level of the virus in their blood after 24 weeks. The investigators also want to understand if the new treatment, MK-8591B, is safe and how well people can handle it.

ELIGIBILITY:
Inclusion:

The main inclusion criteria include but are not limited to the following:

- Has been receiving Bictegravir/Emtricitabine/Tenofovir alafenamide (BIC/FTC/TAF) therapy with documented viral suppression [Human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) <50 copies/mL] for ≥6 months prior to providing documented informed consent and has no history of prior virologic treatment failure on any past or current regimen.

Exclusion:

The main exclusion criteria include but are not limited to the following:

* Has Human immunodeficiency virus type 2 (HIV-2) infection.
* Has a diagnosis of an active Acquired immune deficiency syndrome (AIDS)-defining opportunistic infection.
* Has active hepatitis C virus (HCV) coinfection.
* Has hepatitis B virus (HBV) coinfection.
* Has a history of malignancy ≤5 years prior to providing documented informed consent except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or in situ anal cancer, or cutaneous Kaposi's sarcoma.
* Has prior exposure to Islatravir (ISL) or Ulonivirine (ULO) for any duration any time prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-08-10 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With HIV-1 RNA ≥50 copies/mL at Week 24 | Week 24
  Plasma HIV-1 ribonucleic acid (RNA) quantification will be performed at the central laboratory using a polymerase chain reaction (PCR) assay. Percentage of participants with HIV-1 RNA ≥50 copies/mL will be reported at week 24.
Percentage of Participants who Experience an Adverse Event (AE) | Up to ~ 96 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The percentage of participants who experience an AE will be reported.
Percentage of Participants Discontinuing Study Treatment due to AEs | Up to ~ 96 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The percentage of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Percentage of Participants With HIV-1 RNA ≥50 copies/mL at Week 48 | Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a polymerase chain reaction (PCR) assay. Percentage of participants with HIV-1 RNA ≥50 copies/mL will be reported at week 48.
Percentage of Participants With HIV-1 RNA <50 copies/mL at Week 24 | Week 24
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <50 copies/mL will be reported at week 24.
Percentage of Participants With HIV-1 RNA <50 copies/mL at Week 48 | Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <50 copies/mL will be reported at week 48.
Percentage of Participants With HIV-1 RNA <200 copies/mL at Week 24 | Week 24
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <200 copies/mL will be reported at week 24.
Percentage of Participants With HIV-1 RNA <200 copies/mL at Week 48 | Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <200 copies/mL will be reported at week 48.
Percentage of Participants With HIV-1 RNA ≥50 copies/mL at Week 96 | Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA ≥50 copies/mL will be reported at week 96.
Percentage of Participants With HIV-1 RNA <50 copies/mL at Week 96 | Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <50 copies/mL will be reported at week 96.
Percentage of Participants With HIV-1 RNA <200 copies/mL at Week 96 | Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a PCR assay. Percentage of participants with HIV-1 RNA <200 copies/mL will be reported at week 96.
Mean Change From Baseline in CD4+ T-cell Count at Week 24 | Week 24
  The mean change from baseline in CD4+ T-cell count will be calculated at each applicable time point at which CD4+ T-cell count is collected with primary interest at 24 weeks. Blood samples are taken for this purpose. Baseline measurements are defined as the Day 1 value for each participant.
Mean Change From Baseline in CD4+ T-cell Count at Week 48 | Week 48
  The mean change from baseline in CD4+ T-cell count will be calculated at each applicable time point at which CD4+ T-cell count is collected with primary interest at 48 weeks. Blood samples are taken for this purpose. Baseline measurements are defined as the Day 1 value for each participant.
Mean Change From Baseline in CD4+ T-cell Count at Week 96 | Week 96
  The mean change from baseline in CD4+ T-cell count will be calculated at each applicable time point at which CD4+ T-cell count is collected with primary interest at 96 weeks. Blood samples are taken for this purpose. Baseline measurements are defined as the Day 1 value for each participant.
Percentage of Participants With Development of Viral Drug Resistance to any Component of Study Intervention at Week 24 | Week 24
  Antiviral drug resistance is the reduced susceptibility of the virus to the study intervention. Participants with HIV-1 RNA ≥400 copies/mL will be included in the resistance analyses. Participants who have test results showing signs of viral resistance will also be included for analysis, irrespective of the viral load. Percentage of participants in each treatment group who have evidence of resistance-associated substitutions will be analyzed at week 24.
Percentage of Participants With Development of Viral Drug Resistance to any Component of Study Intervention at Week 48 | Week 48
  Antiviral drug resistance is the reduced susceptibility of the virus to the study intervention. Participants with HIV-1 RNA ≥400 copies/mL will be included in the resistance analyses. Participants who have test results showing signs of viral resistance will also be included for analysis, irrespective of the viral load. Percentage of participants in each treatment group who have evidence of resistance-associated substitutions will be analyzed at week 48.
Percentage of Participants With Development of Viral Drug Resistance to any Component of Study Intervention at Week 96 | Week 96
  Antiviral drug resistance is the reduced susceptibility of the virus to the study intervention. Participants with HIV-1 RNA ≥400 copies/mL will be included in the resistance analyses. Participants who have test results showing signs of viral resistance will also be included for analysis, irrespective of the viral load. Percentage of participants in each treatment group who have evidence of resistance-associated substitutions will be analyzed at week 96.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (23):
- United States (11):
  - Zuckerberg San Francisco General Hospital and Trauma Center ( Site 4107), San Francisco, California
  - Mills Clinical Research ( Site 4109), West Hollywood, California
  - Georgetown University Medical Center ( Site 4106), Washington D.C., District of Columbia
  - Orlando Immunology Center ( Site 4103), Orlando, Florida
  - Triple O Research Institute ( Site 4111), West Palm Beach, Florida
  - Chatham County Health Department - Chatham CARE Center ( Site 4116), Savannah, Georgia
  - KC CARE Health Center ( Site 4101), Kansas City, Missouri
  - Regional Center for Infectious Diseases ( Site 4115), Greensboro, North Carolina
  - Central Texas Clinical Research ( Site 4100), Austin, Texas
  - Prism Health North Texas, Oak Cliff Health Center ( Site 4114), Dallas, Texas
  - DCOL Center for Clinical Research ( Site 4112), Longview, Texas
- Australia (5):
  - Momentum Clinical Research - Darlinghurst ( Site 4260), Darlinghurst, New South Wales
  - St. Vincent's Hospital ( Site 4263), Darlinghurst, New South Wales
  - Momentum Clinical Research Fortitude Valley ( Site 4261), Fortitude Valley, Queensland
  - The Alfred Hospital ( Site 4264), Melbourne, Victoria
  - Prahran Market Clinic ( Site 4262), Prahran, Victoria
- Puerto Rico (3):
  - Ponce Medical School Foundation Inc./CAIMED Center ( Site 4301), Ponce
  - Clinical Research Puerto Rico ( Site 4300), San Juan
  - HOPE Clinical Research ( Site 4303), San Juan
- Switzerland (4):
  - University Hospital Basel-Infectiology ( Site 4402), Basel, Canton of Basel-City
  - Inselspital Bern-Inselspital Infektiologie ( Site 4403), Bern, Canton of Bern
  - Hôpitaux Universitaires de Genève (HUG)-Infectious Disease Department ( Site 4404), Geneva, Canton of Geneva
  - Ospedale Regionale di Lugano, Sede Civico-Servizio Malattie Infettive ( Site 4405), Lugano, Canton Ticino

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com